CLINICAL TRIAL: NCT06129578
Title: Plant Protein Supplementation Within a Healthy Lifestyle Modulates Plasma Circulating Amino Acids and Improves the Health Status of Overweight Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sergio Montserrat de la Paz (Other)
Collaborators: Spanish National Research Council (Other Government)
Responsible Party: Sponsor-Investigator, Sergio Montserrat de la Paz, Professor, University of Seville
Organization: University of Seville (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 2246-N-20
Record Dates: First submitted 2023-11-02; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Obesity; Metabolic Syndrome; Metabolic Disorder; Inflammation; Immune System and Related Disorders
MeSH Terms: conditions — Obesity; Metabolic Syndrome; Metabolic Diseases; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: Mediterranean diet supplement with 20 g / day of hemp protein. — All participants followed a low-energy diet (1315 kcal/daily) based on Mediterranean diet for 12 weeks, supplement with 20 g / day of hemp protein. The specific menu was designed by a trainee nutritionist. The program prescribed five meals a day, with the time customized to fit the lifestyle of each patient. Based on the baseline metabolism, the energy and nutritional parameters of every patient were computed. Patients reported the dietary intake data daily.
  The intervention included face to face visit every two weeks, individual nutrition counseling and education sessions.

SUMMARY:
A dietary pattern based on Mediterranean diet has been reported as healthy for humans, as well as doing aerobic exercise regularly, diminishing the development of potential inflammation in subjects. Protein intake has been proposed as nutritional strategy to further improve these positives outcomes in terms of preventing inflammation diseases. In this work, overweight patients followed a Mediterranean diet together with aerobic exercise according to WHO-guidelines and were supplemented with 20 g of hemp protein/day, for twelve weeks.

Anthropometric and biochemical measures (including analysis of oligoelements), as well as plasma circulating amino acids were evaluated in each patient at the end of the intervention, to assess whether biologically relevant changes could be observed.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 65 years old
* waist circumference ≥94cm in men and ≥88cm in women
* MET<4

Exclusion Criteria:

* prediabetic patients on pharmacotherapy
* subjects suffering from medical issues (e.g., diabetes or another chronic disease)
* smokers
* pregnant or lactating women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Evolution of cytokines in intervention | [Time Frame: Up to 6 hours]
  Pro-inflammatory and anti-inflammatory cytokines, including NFα, IL-1β, IL-6, IL-8, IL-10, ICAM-1, MCP-1, leptin, and adiponectin, in plasma will be measured using appropriate methods (EIA, ELISA, and/or Bioplex multiplex system) (mg/dl).
Effect of the intervention on subjects' biochemical measures | [Time Frame: Up to 6 hours]
  Total cholesterol and triglycerides (TAG) (mg/dL) were determined by enzymatic methods (CHOD-PAP and GPO-PAP, respectively; Roche Diagnostics, Basel, Switzerland). High density lipoprotein-cholesterol (HDL-C) (mg/dL= was determined after precipitation with phosphotungstic acid. Low-density lipoprotein cholesterol (LDL-C) (mg/dL) was calculated with the Firedewald formula. Blood glucose levels, measured by biochemical procedures (mg/dL).
Effect of the intervention on the serum amino acid levels of the subjects. | [Time Frame: Up to 6 hours]
  The amino acid content in plasma (μmol/L) samples analyses were carried out in the University of Sevilla (General Microanalysis Research Service), using an amino acid analyzer BIOCHROM 30, following an amino acid analysis method based on ion exchange chromatography with post column derivatization with ninhydrin.
Effect of the intervention on the serum mineral levels of the subjects. | [Time Frame: Up to 6 hours]
  Mineral content (μgl/L) was evaluated using UV or colorimetrics commercial kits (Bioscience Medical).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Seville, Seville, Spain

IPD SHARING:
Plan to Share IPD: Undecided